CLINICAL TRIAL: NCT02795845
Title: Oral Probiotics for the Treatment and Prevention of Vulvovaginal Infections in Pregnancy - Double-blind, Randomized, Placebo-controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0079-15
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2021-08

CONDITIONS: Bacterial Vaginosis and Vaginal Candidiasis At Pregnancy
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Primary prevention- probiotic capsules (Experimental): patients with normal vaginal flora in the experimental arm will be treated with Probiotic capsules (containing L. acidophilus, L. Paracasei, L. Rhamnosus, streptococcus thermophilus, Bifidobacterium bifidum and B. Lactis).
  one capsule twice a day until delivery.
  Interventions: Dietary Supplement: Probiotic Capsule containing L. acidophilus, L. Paracasei, L. Rhamnosus, streptococcus thermophilus and Bifidobacterium bifidum
- Primary prevention - Placebo (Placebo Comparator): patients with normal vaginal flora in the placebo arm will be treated with a capsule without active ingredient, one capsule twice a day until delivery.
  Interventions: Other: Placebo
- Secondary prevention - probiotic capsules (Experimental): Patients with abnormal vaginal flora/bacterial vaginosis or vaginal candidiasis in the experimental arm will be treated with antibiotic (either clindamycin, metronidazole or both if necessary) or antimycotic treatment. Once the infection was eradicated, the patient will be given probiotic capsules.
  Interventions: Dietary Supplement: Probiotic Capsule containing L. acidophilus, L. Paracasei, L. Rhamnosus, streptococcus thermophilus and Bifidobacterium bifidum
- Secondary prevention - Placebo (Placebo Comparator): Patients with abnormal vaginal flora/bacterial vaginosis or vaginal candidiasis in the experimental arm will be treated with antibiotic (either clindamycin, metronidazole or both if necessary) or antimycotic treatment. Once the infection was eradicated, the patient will be given placebo without active ingredient.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Capsule containing L. acidophilus, L. Paracasei, L. Rhamnosus, streptococcus thermophilus and Bifidobacterium bifidum — Probiotic
  Arms: Primary prevention- probiotic capsules; Secondary prevention - probiotic capsules
Other: Placebo — capsule without active ingredient
  Arms: Primary prevention - Placebo; Secondary prevention - Placebo

SUMMARY:
During pregnancy, bacterial vaginosis (BV), abnormal vaginal flora (AVF) and vulvovaginal candidiasis (VVC) are associated with serious complications and discomfort. Yet, treatment options are limited. Lactobacilli administration was suggested to treat and prevent vaginal infections. However, this has not been examined in pregnant women, the information regarding oral treatment is scarce, and the mechanisms in which oral ingestion of probiotics induce vaginal lactobacilli proliferation are not well established. In the present study we will examine if oral probiotics are effective in prevention of vaginal infections by migration of lactobacilli from the digestive system to the vagina in pregnant women.

DETAILED DESCRIPTION:
During pregnancy, bacterial vaginosis (BV), abnormal vaginal flora (AVF) and vulvovaginal candidiasis (VVC) are associated with serious complications and discomfort. Yet, treatment options are limited. Lactobacilli administration was suggested to treat and prevent vaginal infections. However, this has not been examined in pregnant women, the information regarding oral treatment is scarce, and the mechanisms in which oral ingestion of probiotics induce vaginal lactobacilli proliferation are not well established.

Working hypothesis: Oral probiotics will be effective in prevention of vaginal infections by migration of lactobacilli from the digestive system to the vagina in pregnant women.

Type of research and methods of data collection: randomized placebo-controlled trial.

Pregnant patients with symptoms consisted with vaginal infection will be examined and vaginal smear will be obtained, according to which the patients will be allocated to the following groups:

Primary prevention - women with normal vaginal flora Secondary prevention - women positive for AVF/BV and/or VVC- those women will be treated with antibiotic and/or antimycotic treatment. Following treatment, another smear will be taken to confirm infection eradication. If infection is still present, additional antibiotic and/or antimycotic treatment will be administered after which additional smear will be taken. Women with normal vaginal flora (after one of two treatments) will be recruited for the secondary prevention group.

In each group the patients will be divided into two subgroups, which will receive one capsule twice a day of either the Probiotic Femina ׀׀ capsules or placebo.

At the initial examination and once a month all the study groups will be tested for the presence of AVF/BV and candida. Additional vaginal samples will be taken to evaluate the presence of lactobacilli from the capsule and semi-quantitative assessment of vaginal lactobacilli.

ELIGIBILITY:
Inclusion criteria:

1. Women who will report on vaginal discharge or signs/symptoms consistent with vaginal/vulvar infection
2. Above 18 years old
3. pregnant women until 30th weeks of gestation
4. Willing to participate and singed on consent form

Exclusion criteria:

1. Patient refuse to participate in the study
2. Women with preterm premature rupture of the membranes (at enrollment)
3. Immunocompromised women (e.g. autoimmune diseases treated medically)
4. Failure to eradicate BV/AVF and/or VVC after 2 treatment cycles
5. Trichomonas infection at enrollment
6. Allergy to Soy (The capsules are manufactured in same line as Soy and fish therefore may contain those allergens)
7. Allergy to Fish (The capsules are manufactured in same line as Soy and fish therefore may contain those allergens)
8. Women who take probiotic treatment orally or vaginally that refuse to discontinue treatment.
9. Vaginal swab result suitable for study arm in which enrollment was completed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
The degree of vaginal lactobacilli colonization in the probiotic formula group versus placebo | Around 4 months
  Lactobacilli culture will be made from a vaginal specimen. The pattern of bacterial growth will be used for a semi-quantitative interpretation in a scale of 0-no vaginal colonization to 4-substantial colonization.
The rate of women in the primary prevention group, who developed any vaginal infection (BV/AVF/VVC) during the study period until delivery in the probiotic formula group versus placebo. | From date of randomization until the date of first documented episode or until delivery (around 4 months)
The rate of women in the second prevention group who developed any vaginal infection (BV/AVF/VVC) during the study period until delivery in the probiotic formula group versus placebo. | Until delivery (around 4 months)

SECONDARY OUTCOMES:
Duration of time from the beginning of the study until an episode of vaginal infection (either AVF/BV or VVC). | From randomization until delivery (around 4 months)
The number of episodes of vaginal infections during pregnancy (either AVF/BV or VVC). | From randomization until delivery (around 4 months)
The rate of women, who suffer from obstetrical complications | From randomization until delivery (around 4 months)
  preterm labor, intrauterine growth restriction (IUGR), PPROM, chorioamnionitis, post-partum fever, post-partum endometritis
The rate and type of adverse effects in the probiotic versus placebo groups (e.g gastrointestinal symptoms). | From randomization until two weeks after delivery (around 4 months)
Number of urinary tract infections during the study period | From randomization until delivery (around 4 months)
The rate of neonatal complications | 30 days after delivery
  Neonatal acute respiratory distress syndrome, intraventricular hemorrhage, neonatal sepsis, admission to the neonatal intensive care unit
The rate of women in the primary prevention group who developed AVF/BV during the study period until delivery in the probiotic formula group versus placebo. | From randomization until delivery (around 4 months)
The rate of women in the primary prevention group who developed VVC during the study period until delivery in the probiotic formula group versus placebo. | From randomization until delivery (around 4 months)
The rate of women in the second prevention group who developed AVF/BV during the study period until delivery in the probiotic formula group versus placebo. | From randomization until delivery (around 4 months)
The rate of women in the second prevention group who developed VVC during the study period until delivery in the probiotic formula group versus placebo. | From randomization until delivery (around 4 months)

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Departement of obstetric and gynecology, HaEmek medical center, Afula
  - Women Helth center - Clalit, Afula
  - The holy family hospital, Nazareth

IPD SHARING:
Plan to Share IPD: No